CLINICAL TRIAL: NCT03178591
Title: Effects of DPP4 Inhibitor Versus SGLT2 Inhibitor on Ischemic Burden in Stable Ischemic Heart Disease Patients
Brief Title: Effects of DPP4 Inhibitor Versus SGLT2 Inhibitor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Arintaya Phrommintikul, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-2559-04116
Record Dates: First submitted 2017-01-09; First posted 2017-06-07 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2; Ischemic Heart Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Ischemia | interventions — Vildagliptin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vildagliptin (Active Comparator): Vildagliptin is a dipeptidyl peptidase-4 inhibitor (DPP-4 inhibitor) Dose of Vildagliptin is 50 mg once or twice daily.
  Interventions: Drug: vildagliptin
- Dapagliflozin (Active Comparator): Dapagliflozin is a sodium glucose cotransporter-2 (SGLT-2 inhibitor) Dose of Dapagliflozin is 10 mg once daily.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: vildagliptin
  Arms: vildagliptin
Drug: Dapagliflozin
  Arms: Dapagliflozin

SUMMARY:
Type 2 diabetes mellitus (type 2 DM) is an important disease with increasing prevalence worldwide. More than 60% of diabetes patients die of CVD. Diabetes is associated with 2-to 4- fold increase in the risk of coronary artery disease (CAD). Diabetes patients with stable ischemic heart disease may have more prevalent of asymptomatic ischemia or silent ischemia due to autonomic neuropathy. Therefore, detection of total myocardial ischemia including both symptomatic and silent ischemia using ambulatory electrocardiogram monitoring may provide better accuracy in ischemic burden and prognosis in diabetes patients. DDP-4 inhibitors have favorable effects on atherosclerotic risk factors beyond glycemic control. Furthermore, DPP-4 inhibitors may have favorable effects on ischemic preconditioning in patients with CAD. For this study we aim to compare the effects of between vildagliptin and Dapagliflozin on ischemic burden defined by total ischemic time, markers of autonomic function, biomarkers of myocardial injury and biomarkers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age > 21), male or non-child bearing potential female
2. Inadequately controlled type 2 diabetes with at least half maximum dose of metformin (HbA1C > 6.5 and < 9.0%)
3. Stable documented CAD defined as the followings:

   1. Stable angina with > 70% stenosis of at least one major epicardial artery from coronary angiogram (CAG) or coronary CTA
   2. Post myocardial infarction (> 30 days)

Exclusion Criteria:

1. Significant renal function (eGFR < 30ml/min)
2. Significant hepatic impairment or ALT/AST elevations beyond X2 upper normal limit or known hepatic failure
3. Planned coronary intervention or planed surgical intervention (PCI or CABG)
4. Recent (<30 day) acute coronary syndrome (ACS)
5. Hypersensitivity to either of the study drug components
6. History of lactic acidosis
7. Type 1 diabetes
8. Current HbA1c >9%
9. Current Insulin treatment
10. Active treatment with GLP-1 or other DPP4i medication
11. Inability to comply with study protocol
12. Active malignancy other than basal cell carcinoma
13. Clinically advanced congestive heart failure - NYHA III-IV
14. Severe left ventricular dysfunction (LVEF<25%)
15. Recent heart failure decompensation (<3 months)
16. Chronic inflammation (i.e. inflammatory bowel disease, lupus, inflammatory arthritis, rheumatoid arthritis) or chronic infection (i.e. chronic diabetic foot infection)
17. Pregnancy, lactation or child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of participants who has ST segment depression in ambulatory ECG monitoring during 24 hours at 6 months between DPP4 inhibitor (vildaglptin) group and SGLT2 inhibitors (Dapagliflozin) group | 6 months
Number of myocardial dysfunction which verified by Exercise stress test at 6 month between DPP4 inhibitor (vildaglptin) group and SGLT2 inhibitors (Dapagliflozin) group | 6 months
The event of autonomic dysfunction from heart rate variability, heart rate turbulence, QT interval at 6 month between DPP4 inhibitor (vildaglptin) group and SGLT2 inhibitors (Dapagliflozin) group | 6 months
The myocardial injury event which verified by hsTnT level at 6 month between DPP4 inhibitor (vildaglptin) group and SGLT2 inhibitors (Dapagliflozin) group | 6 months
The inflammation event which verified by hsCRP, IL-6 and TNF-alpha level at 6 month between DPP4 inhibitor (vildaglptin) group and SGLT2 inhibitors (Dapagliflozin) group | 6 months
The oxidative stress event which verified by MDA and 8-isoprostaglandin F2 alpha level at 6 month between DPP4 inhibitor (vildaglptin) group and SGLT2 inhibitors (Dapagliflozin) group | 6 months
The ventricular wall stretch event which verified by N-terminal ProBNP level between DPP4 inhibitor (vildaglptin) group and SGLT2 inhibitors (Dapagliflozin) group. | 6 months
The average of systolic blood pressure at 6 month between DPP4 inhibitor (vildaglptin) group and SGLT2 inhibitors (Dapagliflozin) group. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arintaya Phrommintikul, MD, Study Chair — Faculty of Medicine, Chiang Mai University
Locations (1):
- Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand